CLINICAL TRIAL: NCT01600911
Title: Establish a Vegetable Signature Database From Human Metabolomics Responses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC0991003
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Human Metabolomic Responses to Plant Foods; Blood Pressure
Keywords: metabolomics; nutri-metabolomics; plant food; blood pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Low phytochemical diet(LPD), high phytochemical diet(HPD) — LPD is a basal diet which low in soy,vegetable and fruit and other plant food to approach low phytochemical. HPD is the diet which add two serving test vegetable in the lunch of LPD.

SUMMARY:
Vegetable is well known to prevent chronic disease,however, the mechanism of its nutrients and non-nutrients still remains to be discovered.We design a feeding study which provides plant foods to subjects one by another and monitoring metabolomic changes up to 7 hours.The goal of this study is to establish a protocol for documenting metabolomics response to plant foods and try to characterize plant foods in terms of their anti-hypertension potentials with metabolomic profiling information.

ELIGIBILITY:
Inclusion Criteria:

* Age :18-60 years
* Body Mass Index :18.5-30(kg/m2)
* Non-smoking,alcohol abusing,and other bad hobbies

Exclusion Criteria:

* With regular drug intake e.g. anti-hypertensive or antidiabetes drug or history of immune, hepatic and metabolic disease or other unsuitable disorders e.g. cancer.
* unwilling to stop regular food supplement e.g. vitamins, herb
* cannot cooperate with designed diet
* History of urinary tract infection or antibiotic use within the previous 3 month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure | one day
  fasting, before lunch,and every 1 hr after lunch

SECONDARY OUTCOMES:
metabolomic profile of serum and urine | one day
  serum sample will be measure fasting ,before lunch,and every 1 hr after lunch;urine sample will be measure fasting ,before lunch(0hr),0-2 hr,2-4hr 4-7hr after lunch

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- National Health Research institues, Taiwan, Miaoli County, Taiwan